CLINICAL TRIAL: NCT02252016
Title: A Phase III Double Blind Clinical Trial to Study the Efficacy and Safety of the Combination Regimen of MK-5172 and MK-8742 in Subjects With Chronic HCV GT1, GT4 and GT6 Infection With Inherited Blood Disorders With and Without HIV Co-Infection
Brief Title: Grazoprevir (MK-5172) and Elbasvir (MK-8742) Combination for Chronic Hepatitis C Virus (HCV) Genotypes 1, 4, and 6 (MK-5172-065)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5172-065; 2014-002356-27 (EudraCT Number)
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Results first posted 2017-01-19 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-09

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — elbasvir-grazoprevir drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate Treatment (Experimental): Participants will take grazoprevir 100 mg + elbasvir 50 mg once daily during the 12-week treatment period and then will be monitored for safety during a 24-week follow-up period.
  Interventions: Drug: Grazoprevir + Elbasvir
- Deferred Treatment (Placebo Comparator): Participants will take placebo tablets once daily during the 12-week treatment period and will then be monitored for safety during a 4-week follow-up period. Participants will then begin open-label treatment with grazoprevir 100 mg + elbasvir 50 mg for a 12-week treatment period and will then be monitored for safety during a 24-week follow-up period.
  Interventions: Drug: Grazoprevir + Elbasvir; Drug: Placebo

INTERVENTIONS:
Drug: Grazoprevir + Elbasvir — FDC tablet containing grazoprevir 100 mg + elbasvir 50 mg taken once daily by mouth.
Drug: Placebo — Placebo tablets matching grazoprevir + elbasvir FDC tablets taken once daily by mouth.
  Arms: Deferred Treatment

SUMMARY:
This is a randomized, multi-site, placebo-controlled trial of a fixed dose combination (FDC) of grazoprevir (MK-5172) 100 mg + elbasvir (MK-8742) 50 mg in participants with chronic Hepatitis C Virus (HCV) genotype (GT) 1, GT4 or GT6 with inherited blood disorders. The primary hypothesis is that the proportion of participants treated with grazoprevir+elbasvir achieving Sustained Virologic Response (SVR) 12 weeks after the end of all study therapy (SVR12) will be greater than the reference rate of 40%.

ELIGIBILITY:
Inclusion Criteria:

* has HCV GT1, GT4, or GT6 with sickle cell anemia, thalassemia, or hemophilia/von Willebrand disease
* has cirrhosis or is non-cirrhotic
* is human immunodeficiency virus (HIV) coinfected or not infected with HIV
* is a female of non childbearing potential, or is male or female and uses an acceptable method(s) of contraception

Exclusion Criteria:

* has evidence of decompensated liver disease
* is coinfected with hepatitis B
* has had a malignancy ≤5 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer
* has hepatocellular carcinoma (HCC) or is under evaluation for HCC
* has clinically-relevant drug or alcohol abuse within 12 months of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2014-10-22 (Actual); Primary Completion 2015-12-07 (Actual); Study Completion 2016-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Hezode C, Colombo M, Bourliere M, Spengler U, Ben-Ari Z, Strasser SI, Lee WM, Morgan L, Qiu J, Hwang P, Robertson M, Nguyen BY, Barr E, Wahl J, Haber B, Chase R, Talwani R, Marco VD; C-EDGE IBLD Study Investigators. Elbasvir/Grazoprevir for Patients With Hepatitis C Virus Infection and Inherited Blood Disorders: A Phase III Study. Hepatology. 2017 Sep;66(3):736-745. doi: 10.1002/hep.29139. Epub 2017 Jul 20. PMID 28256747
- [Derived] Asselah T, Reesink H, Gerstoft J, de Ledinghen V, Pockros PJ, Robertson M, Hwang P, Asante-Appiah E, Wahl J, Nguyen BY, Barr E, Talwani R, Serfaty L. Efficacy of elbasvir and grazoprevir in participants with hepatitis C virus genotype 4 infection: A pooled analysis. Liver Int. 2018 Sep;38(9):1583-1591. doi: 10.1111/liv.13727. Epub 2018 Mar 31. PMID 29461687

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult participants with hepatitis C virus (HCV) genotypes (GT)1, GT4, and GT6 with inherited blood disorders and with or without human immunodeficiency virus (HIV) co-infection were recruited at study centers around the world.
Groups:
- Immediate Treatment: Participants took grazoprevir 100 mg + elbasvir 50 mg once daily (q.d.) during the initial 12-week treatment period, followed by a 24-week safety monitoring period.
- Deferred Treatment: Participants took placebo tablets q.d. during the initial 12-week treatment period, and then underwent a 4-week safety monitoring follow-up period. Next, participants took open-label grazoprevir 100 mg + elbasvir 50 mg q.d. for 12 weeks, followed by a 24-week safety monitoring period.
Period: Overall Study
Arm/Group | Immediate Treatment | Deferred Treatment
Started | 107 | 52
Completed | 104 (Completed = completed 24 weeks of follow-up) | 49 (Completed = completed 24 weeks of follow-up)
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 2 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Treatment | Deferred Treatment | Total
Number analyzed (Participants) | 107 | 52 | 159
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.2 (11.2) | 42.5 (9.8) | 43.6 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 13 | 40
  Male | 80 | 39 | 119

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Virologic Response 12 Weeks After Completing Study Therapy (SVR12)
Description: The percentage of participants in the both arms achieving SVR12 (i.e., HCV riboncleic acid [RNA] level below the lower limit of quantification [LLoQ] 12 weeks after completing study therapy) was determined. HCV RNA levels were measured using the Roche COBAS™ Taqman™ HCV Test v2.0 (High Pure System), which has a LLoQ of <15 IU/mL.
Time Frame: 12 weeks after completing study therapy (Week 24)
Population: The Full Analysis Set (FAS) consists of all treated participants in both arms other than those who discontinued with reasons unrelated to the treatment regimen or HCV response.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Immediate Treatment | Deferred Treatment
Number analyzed (Participants) | 107 | 49
Percentage of participants | 93.5 [87.0 to 97.3] | 91.8 [80.4 to 97.7]

2. Primary Outcome: Percentage of Participants Experiencing an Adverse Event (AE)
Description: An AE is any untoward medical occurrence which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to Week 14
Population: The All-Participants-as-Treated (APaT) population includes all participants receiving ≥1 dose(s) of study drug. For the Deferred Treatment arm, data indicate results obtained during the initial 12-week placebo treatment period.
Measure: Number; unit: Percentage of Participants
Arm/Group | Immediate Treatment | Deferred Treatment
Number analyzed (Participants) | 107 | 52
Percentage of Participants | 72.9 | 65.4
Statistical Analysis 1: Comparison: Immediate Treatment vs Deferred Treatment; The estimated difference (± 95% confidence interval [CI]) in percentage of participants experiencing an AE in the Immediate versus Deferred arms was determined; Test type: Superiority or Other; Mean Difference (Final Values) = 7.5, 95% CI 2-sided [-7.3 to 23.3]

3. Primary Outcome: Percentage of Participants Discontinuing From Study Treatment Due to an AE(s)
Description: as for outcome 2
Time Frame: Up to Week 12
Population: The APaT population includes all participants receiving ≥1 dose(s) of study drug. For the Deferred Treatment arm, data indicate results obtained during the initial 12-week placebo treatment period.
Measure: Number; unit: Percentage of Participants
Arm/Group | Immediate Treatment | Deferred Treatment
Number analyzed (Participants) | 107 | 52
Percentage of Participants | 0.0 | 1.9
Statistical Analysis 1: Comparison: Immediate Treatment; The estimated difference (± 95% CI) in percentage of participants withdrawing from study treatment due to an AE(s) in the Immediate versus Deferred arms was determined; Test type: Superiority or Other; p = 0.155, Miettinen & Nurminen method; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-10.2 to 1.6]

4. Secondary Outcome: Percentage of Participants Achieving Sustained Virologic Response 24 Weeks After Completing Study Therapy (SVR24)
Description: The percentage of participants in both arms achieving SVR24 (i.e., HCV RNA level below the LLoQ 24 weeks after completing study therapy) was determined. HCV RNA levels were measured using the Roche COBAS™ Taqman™ HCV Test v2.0 (High Pure System), which has a LLoQ of <15 IU/mL.
Time Frame: 24 weeks after completing study therapy (Week 36)
Population: The FAS consists of all treated participants in both arms other than those who discontinued with reasons unrelated to the treatment regimen or HCV response.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Immediate Treatment | Deferred Treatment
Number analyzed (Participants) | 107 | 49
Percentage of participants | 90.7 [83.5 to 95.4] | 91.8 [80.4 to 97.7]

ADVERSE EVENTS:
Time Frame: Up to 52 weeks
Description: An AE is any untoward medical occurrence which does not necessarily have to have a causal relationship with this treatment. AEs were reported for all participants receiving ≥ 1 dose of study treatment.
Groups:
- Deferred Treatment: Placebo Phase: Participants took placebo tablets q.d. during the initial 12-week treatment period, and then underwent a 4-week safety monitoring follow-up period. Next, participants took open-label grazoprevir 100 mg + elbasvir 50 mg q.d. for 12 weeks, followed by a 24-week safety monitoring period.
Arm/Group | Immediate Treatment | Deferred Treatment: Placebo Phase
Serious Adverse Events (participants affected / at risk) | 6/107 | 6/52
Other Adverse Events (participants affected / at risk) | 78/107 | 34/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Immediate Treatment (N=107) | Deferred Treatment: Placebo Phase (N=52)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 1 | 2
Myocardial infarction (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Immediate Treatment (N=107) | Deferred Treatment: Placebo Phase (N=52)
Abdominal distension (Gastrointestinal disorders) | 2 | 3
Abdominal pain (Gastrointestinal disorders) | 7 | 2
Diarrhoea (Gastrointestinal disorders) | 4 | 3
Nausea (Gastrointestinal disorders) | 9 | 8
Asthenia (General disorders) | 8 | 2
Fatigue (General disorders) | 18 | 4
Pyrexia (General disorders) | 6 | 0
Nasopharyngitis (Infections and infestations) | 6 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 3
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 3 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 4
Headache (Nervous system disorders) | 23 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation.